CLINICAL TRIAL: NCT03928028
Title: Shifting Perspectives: Enhancing Outcomes in Adolescent Anorexia Nervosa With Cognitive Remediation Therapy (CRT)
Brief Title: Shifting Perspectives: Enhancing Outcomes in Anorexia Nervosa With CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 19-016064; 1R61MH119262-01 (NIH)
Record Dates: First submitted 2019-04-08; First posted 2019-04-25 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Random assignment to one of three groups.
Who Masked: Outcomes Assessor
Masking Description: Any study team member who is assessing for outcomes will not which participant/family is in which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Family Based Treatment (FBT) (Active Comparator): Families will receive 15 sessions of FBT alone.
  Interventions: Behavioral: Family Based Treatment
- FBT w/ Parent-focused Cognitive Remediation Therapy (Experimental): Family Based Treatment with Parent-focused Cognitive Remediation Therapy (CRT): Families will receive 15 sessions of parent focused CRT followed Family Based Treatment over six months.
  Interventions: Behavioral: Cognitive Remediation Therapy; Behavioral: Family Based Treatment
- FBT w/Adolescent-focused Cognitive Remediation Therapy (Experimental): Family Based Treatment with Adolescent-focused Cognitive Remediation Therapy (CRT): Families will receive 15 sessions of adolescent focused CRT followed by Family Based Treatment over six months.
  Interventions: Behavioral: Cognitive Remediation Therapy; Behavioral: Family Based Treatment

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — Cognitive Remediation Therapy (CRT) is an adjunctive treatment focused on increasing set-shifting ability and developing meta-cognition.
  Other Names: CRT
  Arms: FBT w/ Parent-focused Cognitive Remediation Therapy; FBT w/Adolescent-focused Cognitive Remediation Therapy
Behavioral: Family Based Treatment — Family Based Treatment (FBT) is an evidence based treatment in which parents are responsible for adolescent re-nourishment. They play an active role in treatment and their self-efficacy to make decisions regarding their child's treatment is empowered.
  Other Names: FBT

SUMMARY:
Anorexia Nervosa is a serious life-threatening illness with a typical age of onset in adolescence; if not effectively treated, it has the potential to significantly impact adolescent development and quality of life. Research on executive functioning in anorexia nervosa indicates that it may be a viable target for intervention that could improve outcome. The current project focuses on determining whether or not the investigators can improve set-shifting in parents and affected adolescents in the hopes that improvements in set-shifting will, ultimately, improve outcome.

DETAILED DESCRIPTION:
This application seeks support for a phased project. In the initial (R61) 2-year phase, the investigators will establish that Cognitive Remediation Therapy (CRT) can increase set-shifting in parents of and/or adolescents with Anorexia Nervosa (AN). The second aim is to determine the appropriate dose needed to achieve positive change in set-shifting. Attaining this milestone would trigger support for three additional years (R33) to confirm target engagement and appropriate dose. The investigators will also evaluate whether or not adding CRT to Family Based Treatment (FBT) will improve outcome compared to FBT alone. Set-shifting (a type of executive functioning often referred to as cognitive flexibility) inefficiencies are hypothesized to be an endophenotype of AN and are, therefore, heritable. Cognitive flexibility can be impacted negatively by situational factors such as malnutrition, stress, and anxiety. It is likely that both adolescents (who are malnourished) and parents (who are under stress) experience significant state-based reduction in their cognitive flexibility during AN and its treatment. While cognitive flexibility can be increased through CRT, there is a significant gap in the knowledge about how to apply CRT to the treatment of adolescent AN, specifically concerning the most appropriate target for CRT: parents or adolescents? The majority of research on CRT with adolescents with AN are pilot and feasibility studies and target set-shifting in adolescents, not parents. The investigators hypothesize that targeting parents may be more impactful for adolescent outcome. First, the investigators must determine if an increase set-shifting via CRT is possible. In the initial R61 phase, the investigators propose to recruit and randomly assign 54 families who have a child with AN to FBT, FBT with parent-focused CRT, or FBT with adolescent-focused CRT. Target engagement will be assessed via neuro-psychological assessment and self-report of cognitive and behavioral flexibility. If the investigators meet these proposed milestones in the R61 phase, they will proceed to the R33 phase. It is possible that one (N = 72 families) or both (N = 93 families) CRT conditions will be examined in the R33 phase. The investigators will confirm the findings from the R61 phase (target engagement and dose of CRT). The investigators will also examine adolescent outcome in FBT alone versus FBT+(parent or adolescent) CRT. They will gather preliminary data on putative moderators and/or mediators across both phases in order to inform results. This phased R61/R33 application is innovative in that it is the first to adapt CRT to parents only. Evidence supporting FBT+CRT to increase set-shifting in parents/adolescents will inform future efforts to leverage understanding of (heritable) neurobiology of AN in adolescents to improve outcome. Further, if CRT for parents significantly improves set-shifting, the investigators can focus efforts on how best to augment current treatments, support parents, and increase positive outcomes for the adolescent and reduce relapse. Even negative results would inform understanding of set-shifting inefficiencies as an endophenotype in AN, its measurement, and usefulness as a target in treatment.

ELIGIBILITY:
Inclusion Criteria:Adolescents

1. Age 12-18
2. Currently meets Diagnostic and Statistical Manual-5 criteria for Anorexia Nervosa
3. Medically stable for outpatient treatment
4. Fluent in English
5. No co-morbid condition that would exclude participation
6. Medical clearance from primary care physician and permission to speak to Primary Care Physician about clinical issues
7. Biological parent or primary caregiver willing to engage in treatment and who live with the adolescent

Inclusion Criteria:Parents

1. Age >18
2. Child with a diagnoses of AN
3. Both parents willing to participate
4. Fluent in English
5. No co-morbid condition that would exclude participation

Exclusion Criteria: Adolescent

1. Adolescent outside age range
2. Adolescent adopted
3. Pregnant adolescent
4. Presence of: pervasive developmental disability, psychosis, bipolar disorder, substance abuse, autism spectrum disorder, or intellectual disability
5. Presence of: a brain disorder or injury (such as TBI) that could impact the ability to engage in treatment
6. Use of anti-psychotic medication
7. Concurrent psychosocial therapy

Exclusion Criteria: Parents

1. Presence of: pervasive developmental disability, psychosis, bipolar disorder, substance abuse, autism spectrum disorder, or intellectual disability.
2. Presence of: a brain disorder or injury (such as TBI) that could impact the ability to engage in treatment
3. Use of anti-psychotic medication

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Alix Timko, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holliday J, Tchanturia K, Landau S, Collier D, Treasure J. Is impaired set-shifting an endophenotype of anorexia nervosa? Am J Psychiatry. 2005 Dec;162(12):2269-75. doi: 10.1176/appi.ajp.162.12.2269. PMID 16330590
- [Background] Lang K, Stahl D, Espie J, Treasure J, Tchanturia K. Set shifting in children and adolescents with anorexia nervosa: an exploratory systematic review and meta-analysis. Int J Eat Disord. 2014 May;47(4):394-9. doi: 10.1002/eat.22235. Epub 2013 Dec 18. PMID 24347025
- [Background] Roberts ME, Tchanturia K, Stahl D, Southgate L, Treasure J. A systematic review and meta-analysis of set-shifting ability in eating disorders. Psychol Med. 2007 Aug;37(8):1075-84. doi: 10.1017/S0033291707009877. Epub 2007 Jan 30. PMID 17261218
- [Background] Roberts ME, Tchanturia K, Treasure JL. Exploring the neurocognitive signature of poor set-shifting in anorexia and bulimia nervosa. J Psychiatr Res. 2010 Oct;44(14):964-70. doi: 10.1016/j.jpsychires.2010.03.001. Epub 2010 Apr 15. PMID 20398910
- [Background] Lang K, Treasure J, Tchanturia K. Is inefficient cognitive processing in anorexia nervosa a familial trait? A neuropsychological pilot study of mothers of offspring with a diagnosis of anorexia nervosa. World J Biol Psychiatry. 2016 Jun;17(4):258-65. doi: 10.3109/15622975.2015.1112035. Epub 2015 Dec 1. PMID 26563611
- [Background] Kucharska K, Kulakowska D, Starzomska M, Rybakowski F, Biernacka K. The improvement in neurocognitive functioning in anorexia nervosa adolescents throughout the integrative model of psychotherapy including cognitive remediation therapy. BMC Psychiatry. 2019 Jan 9;19(1):15. doi: 10.1186/s12888-018-1984-4. PMID 30626367
- [Background] Harrison A, Stavri P, Ormond L, McEnemy F, Akyol D, Qureshi A, Al-Khairulla H. Cognitive remediation therapy for adolescent inpatients with severe and complex anorexia nervosa: A treatment trial. Eur Eat Disord Rev. 2018 May;26(3):230-240. doi: 10.1002/erv.2584. Epub 2018 Mar 15. PMID 29542258
- [Derived] Susanin A, Cooper M, Makara A, Kuschner ES, Timko CA. Autistic characteristics in youth with anorexia nervosa before and after treatment. Eur Eat Disord Rev. 2022 Sep;30(5):664-670. doi: 10.1002/erv.2937. Epub 2022 Jul 3. PMID 35780511
- [Derived] Timko CA, Bhattacharya A, Fitzpatrick KK, Howe H, Rodriguez D, Mears C, Heckert K, Ubel PA, Ehrenreich-May J, Peebles R. The shifting perspectives study protocol: Cognitive remediation therapy as an adjunctive treatment to family based treatment for adolescents with anorexia nervosa. Contemp Clin Trials. 2021 Apr;103:106313. doi: 10.1016/j.cct.2021.106313. Epub 2021 Feb 1. PMID 33539993

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Families
Period: Overall Study
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Started | 63; 21 Families | 57; 19 Families | 57; 19 Families
Mother | 21; 21 Families | 19; 19 Families | 19; 19 Families
Father | 21; 21 Families | 19; 19 Families | 19; 19 Families
Adolescent | 21; 21 Families | 19; 19 Families | 19; 19 Families
Completed | 42; 14 Families | 48; 16 Families | 51; 17 Families
Not Completed | 21; 7 Families | 9; 3 Families | 6; 2 Families
Not completed — Physician Decision | 9 | 6 | 3
Not completed — Withdrawal by Subject | 12 | 3 | 3

BASELINE CHARACTERISTICS:
Population: 59 family units were enrolled. Mothers, Fathers, and adolescents were analyzed separately as groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy | Total
Number analyzed (Participants) | 63 | 57 | 57 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 19 | 19 | 59
  Between 18 and 65 years | 42 | 37 | 38 | 117
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Adolescents, mothers, and fathers are reported separately.
  years
    Adolescents: number analyzed (Participants) | 21 | 19 | 19 | 59
    Adolescents | 15.51 (1.81) | 15.21 (1.53) | 15.25 (1.61) | 15.335 (1.641)
    Mothers: number analyzed (Participants) | 21 | 19 | 19 | 59
    Mothers | 48.18 (3.61) | 47.46 (6.25) | 47.30 (2.997) | 47.66 (4.42)
    Fathers: number analyzed (Participants) | 21 | 19 | 19 | 59
    Fathers | 50.65 (5.98) | 49.93 (6.82) | 48.97 (4.82) | 49.88 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 35 | 110
  Male | 24 | 21 | 22 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 58 | 54 | 55 | 167
  Unknown or Not Reported | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3
  White | 58 | 49 | 53 | 160
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 57 | 57 | 177

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Flexibility - Condition 4 Trail Making Test of DKEFS
Description: The Delis Kaplan Executive Functioning System (D-KEFS) is a standardized assessment of executive functioning normed for ages 8-89 years of age. Raw scores are transformed to scaled scores: the mean is 10 with a standard deviation of 3. Higher scores indicate better performance on the test. Specific sub-tests were chosen to assess inhibitory control and cognitive flexibility. The hypothesis is that Cognitive Remediation Therapy (CRT) will increase flexibility in participants. The D-KEFS was administered at baseline (T1), after 4 weeks (T2), approximately 9 weeks (T3), approximately 17 weeks (T4), and end of treatment (T5). Trail Making Test assesses flexibility in thinking. We use Condition 4 (Number-Letter Switching) to assess flexibility.
Time Frame: 6 months of treatment
Population: All available data is reported for mothers, fathers and adolescents separately. Some data is missing due to COVID-19 impacts on the ability to administer in-person assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Number analyzed (Participants) | 63 | 57 | 57
score on a scale
  Mother- T1: number analyzed (Participants) | 19 | 17 | 17
  Mother- T1 | 11.89 (.875) | 10.94 (2.331) | 11.47 (1.663)
  Mother - T3: number analyzed (Participants) | 14 | 14 | 13
  Mother - T3 | 11.14 (2.742) | 11.86 (2.107) | 12.00 (1.663)
  Mother - T4: number analyzed (Participants) | 11 | 10 | 11
  Mother - T4 | 12.18 (.874) | 12.70 (.675) | 12.27 (1.191)
  1Mother - T5: number analyzed (Participants) | 8 | 9 | 4
  1Mother - T5 | 12.75 (1.165) | 13.11 (.782) | 13.25 (1.708)
  Father - T1: number analyzed (Participants) | 21 | 17 | 17
  Father - T1 | 11.14 (2.265) | 11.06 (1.819) | 11.35 (2.060)
  Father - T3: number analyzed (Participants) | 13 | 14 | 13
  Father - T3 | 11.92 (1.382) | 12.57 (1.342) | 12.23 (1.092)
  Father - T4: number analyzed (Participants) | 11 | 10 | 11
  Father - T4 | 11.82 (2.136) | 13.10 (1.101) | 12.09 (1.640)
  Father - T5: number analyzed (Participants) | 7 | 10 | 6
  Father - T5 | 12.14 (1.069) | 12.80 (.919) | 13.00 (1.549)
  Adolescent - T1: number analyzed (Participants) | 19 | 17 | 17
  Adolescent - T1 | 9.47 (3.151) | 10.59 (2.033) | 10.94 (1.144)
  Adolescent - T3: number analyzed (Participants) | 12 | 14 | 12
  Adolescent - T3 | 9.50 (3.555) | 11.71 (1.773) | 10.83 (1.115)
  Adolescent - T4: number analyzed (Participants) | 10 | 10 | 11
  Adolescent - T4 | 11.00 (2.404) | 12.50 (.850) | 11.64 (1.567)
  Adolescent - T5: number analyzed (Participants) | 8 | 9 | 6
  Adolescent - T5 | 12.50 (1.414) | 12.33 (1.225) | 11.50 (1.643)
Statistical Analysis 1: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares mothers in FBT to mothers in FBT+Parent-focused CRT; Test type: Superiority; p = .507, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 2: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares fathers in FBT to fathers in FBT+Parent-focused CRT; Test type: Superiority; p = .017, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 3: Comparison: Family Based Treatment (FBT) vs FBT w/Adolescent-focused Cognitive Remediation Therapy; This analysis compares adolescents in FBT to adolescents in FBT+Adolescent-focused CRT; Test type: Superiority; p = .139, generalized estimating equation — a priori threshold for statistical significance = .15

2. Primary Outcome: Change in Inhibition - Condition 3 of Color-Word Interference, DKEFS
Description: The Delis Kaplan Executive Functioning System (D-KEFS) is a standardized assessment of executive functioning normed for ages 8-89 years of age. Raw scores are transformed to scaled scores: the mean is 10 with a standard deviation of 3. Higher scores indicate better performance on the test. Specific sub-tests were chosen to assess inhibitory control and cognitive flexibility. The hypothesis is that Cognitive Remediation Therapy (CRT) will increase flexibility in participants. The D-KEFS was administered at baseline (T1), after 4 weeks (T2), approximately 9 weeks (T3), approximately 17 weeks (T4), and end of treatment (T5). Inhibition refers to the ability to inhibit a well learned or salient task in order to do something different; thus, it is related to flexibility. The D-KEFS Color-Word Interference Test (Condition 3: Inhibition) to assess ability to inhibit automatic responses.
Time Frame: 6 months of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Number analyzed (Participants) | 63 | 57 | 57
score on a scale
  Mother -T1: number analyzed (Participants) | 21 | 19 | 19
  Mother -T1 | 11.95 (2.291) | 11.84 (1.608) | 12.21 (2.175)
  Mother - T3: number analyzed (Participants) | 18 | 16 | 18
  Mother - T3 | 12.72 (1.565) | 12.06 (1.237) | 12.94 (2.014)
  Mother - T4: number analyzed (Participants) | 16 | 16 | 17
  Mother - T4 | 13.06 (1.436) | 12.25 (1.528) | 13.12 (1.996)
  Mother - T5: number analyzed (Participants) | 12 | 15 | 15
  Mother - T5 | 13.67 (1.923) | 12.93 (1.668) | 13.33 (1.718)
  Father - T1: number analyzed (Participants) | 21 | 19 | 19
  Father - T1 | 11.14 (2.689) | 12.11 (1.941) | 11.63 (2.52)
  Father - T3: number analyzed (Participants) | 18 | 16 | 18
  Father - T3 | 11.94 (1.798) | 13.06 (1.436) | 12.50 (2.176)
  Father - T4: number analyzed (Participants) | 14 | 16 | 17
  Father - T4 | 12.43 (1.742) | 12.75 (2.840) | 13.00 (1.581)
  Father - T5: number analyzed (Participants) | 11 | 15 | 15
  Father - T5 | 12.55 (1.753) | 13.67 (1.291) | 12.80 (1.740)
  Adolescent-T1: number analyzed (Participants) | 21 | 19 | 18
  Adolescent-T1 | 10.76 (2.300) | 11.95 (2.272) | 11.11 (3.008)
  Adolescent - T3: number analyzed (Participants) | 17 | 16 | 17
  Adolescent - T3 | 11.47 (2.348) | 12.94 (1.482) | 1.35 (2.548)
  Adolescent - T4: number analyzed (Participants) | 15 | 16 | 17
  Adolescent - T4 | 12.67 (1.676) | 13.31 (1.448) | 12.76 (2.412)
  Adolescent - T5: number analyzed (Participants) | 12 | 14 | 15
  Adolescent - T5 | 12.83 (1.642) | 13.14 (1.610) | 13.00 (2.204)
Statistical Analysis 1: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compare mothers in FBT to mothers in FBT+CRTp; Test type: Superiority; p = .389, generalized estimating equation
Statistical Analysis 2: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares fathers in FBT to fathers in FBT+Parent-focused CRT; Test type: Superiority; p = .447, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 3: Comparison: Family Based Treatment (FBT) vs FBT w/Adolescent-focused Cognitive Remediation Therapy; This analysis compares adolescents in FBT to adolescents in FBT+Adolescent-focused CRT; Test type: Superiority; p < .001, generalized estimating equation — a priori threshold for statistical significance = .15

3. Primary Outcome: Change in Cognitive Flexibility - Condition 4 of Color Word Interference of DKEFS
Description: The Delis Kaplan Executive Functioning System (D-KEFS) is a standardized assessment of executive functioning normed for ages 8-89 years of age. Raw scores are transformed to scaled scores: the mean is 10 with a standard deviation of 3. Higher scores indicate better performance on the test. Specific sub-tests were chosen to assess inhibitory control and cognitive flexibility. The hypothesis is that Cognitive Remediation Therapy (CRT) will increase flexibility in participants. The D-KEFS was administered at baseline (T1), after 4 weeks (T2), approximately 9 weeks (T3), approximately 17 weeks (T4), and end of treatment (T5). The D-KEFS Color Word Interference (Condition 4: Inhibition/Switching) assess the ability to switch between alternating rules (a component of set shifting).
Time Frame: 6 months of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Number analyzed (Participants) | 63 | 57 | 57
score on a scale
  Mother - T1: number analyzed (Participants) | 21 | 19 | 19
  Mother - T1 | 11.71 (1.101) | 11.05 (1.615) | 11.95 (2.041)
  Mother - T3: number analyzed (Participants) | 18 | 16 | 18
  Mother - T3 | 12.78 (1.215) | 12.50 (1.633) | 12.78 (1.700)
  Mother - T4: number analyzed (Participants) | 16 | 16 | 17
  Mother - T4 | 12.75 (1.844) | 12.63 (1.586) | 13.35 (1.801)
  Mother - T5: number analyzed (Participants) | 12 | 15 | 15
  Mother - T5 | 13.83 (1.467) | 13.13 (1.356) | 13.40 (1.549)
  Father - T1: number analyzed (Participants) | 21 | 19 | 19
  Father - T1 | 11.67 (2.106) | 12.05 (1.433) | 11.37 (2.929)
  Father - T3: number analyzed (Participants) | 18 | 16 | 18
  Father - T3 | 12.56 (1.504) | 13.13 (1.088) | 12.56 (1.790)
  Father - T4: number analyzed (Participants) | 14 | 16 | 17
  Father - T4 | 12.86 (2.070) | 13.19 (1.515) | 12.94 (1.391)
  Father - T5: number analyzed (Participants) | 11 | 15 | 15
  Father - T5 | 13.09 (1.446) | 13.73 (1.033) | 13.00 (1.414)
  Adolescent - T1: number analyzed (Participants) | 21 | 19 | 18
  Adolescent - T1 | 11.52 (2.994) | 11.63 (2.385) | 11.61 (1.914)
  Adolescent - T3: number analyzed (Participants) | 17 | 16 | 17
  Adolescent - T3 | 12.59 (2.763) | 13.00 (1.751) | 12.35 (2.262)
  Adolescent - T4: number analyzed (Participants) | 15 | 16 | 17
  Adolescent - T4 | 13.60 (1.957) | 13.50 (2.160) | 13.29 (2.114)
  Adolescent - T5: number analyzed (Participants) | 12 | 14 | 15
  Adolescent - T5 | 14.17 (1.030) | 13.71 (2.016) | 13.27 (2.154)
Statistical Analysis 1: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares mothers in FBT to mothers in FBT+Parent-focused CRT; Test type: Superiority; p = .778, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 2: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares mothers in FBT to mothers in FBT+Parent-focused CRT; Test type: Superiority; p = .297, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 3: Comparison: Family Based Treatment (FBT) vs FBT w/Adolescent-focused Cognitive Remediation Therapy; This analysis compares adolescents in FBT to adolescents in FBT+Adolescent-focused CRT; Test type: Superiority; p = .062, generalized estimating equation — a priori threshold for statistical significance = .15

4. Primary Outcome: Change in Cognitive Flexibility - Verbal Fluency Switching of DKEFS
Description: The Delis Kaplan Executive Functioning System (D-KEFS) is a standardized assessment of executive functioning normed for ages 8-89 years of age. Raw scores are transformed to scaled scores: the mean is 10 with a standard deviation of 3. Higher scores indicate better performance on the test. Specific sub-tests were chosen to assess inhibitory control and cognitive flexibility. The hypothesis is that Cognitive Remediation Therapy (CRT) will increase flexibility in participants. The D-KEFS was administered at baseline (T1), after 4 weeks (T2), approximately 9 weeks (T3), approximately 17 weeks (T4), and end of treatment (T5). The D-KEFS Verbal Fluency assesses the ability to shift between concepts. The Switching Correct score is used to assess flexibility.
Time Frame: 6 months of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Number analyzed (Participants) | 63 | 57 | 57
score on a scale
  Mother - T1: number analyzed (Participants) | 20 | 19 | 19
  Mother - T1 | 12.10 (3.478) | 11.95 (2.718) | 11.74 (4.483)
  Mother - T3: number analyzed (Participants) | 19 | 16 | 17
  Mother - T3 | 12.47 (3.717) | 12.44 (3.444) | 11.18 (3.695)
  Mother - T4: number analyzed (Participants) | 16 | 16 | 17
  Mother - T4 | 13.00 (4.195) | 12.44 (3.464) | 13.29 (4.089)
  Mother - T5: number analyzed (Participants) | 12 | 15 | 15
  Mother - T5 | 12.42 (3.288) | 13.53 (2.446) | 13.47 (2.949)
  Father - T1: number analyzed (Participants) | 21 | 19 | 19
  Father - T1 | 11.81 (3.628) | 10.68 (3.973) | 10.63 (3.218)
  Father - T3: number analyzed (Participants) | 19 | 16 | 18
  Father - T3 | 11.68 (3.528) | 11.50 (3.759) | 11.33 (4.102)
  Father - T4: number analyzed (Participants) | 14 | 16 | 16
  Father - T4 | 12.71 (4.286) | 11.88 (3.757) | 12.00 (3.386)
  Father - T5: number analyzed (Participants) | 11 | 14 | 15
  Father - T5 | 12.45 (2.911) | 11.43 (3.694) | 11.73 (4.399)
  Adolescent - T1: number analyzed (Participants) | 20 | 19 | 18
  Adolescent - T1 | 11.55 (3.677) | 12.42 (3.006) | 11.50 (1.917)
  Adolescent - T3: number analyzed (Participants) | 18 | 16 | 17
  Adolescent - T3 | 10.89 (3.411) | 12.31 (3.135) | 9.88 (3.967)
  Adolescent - T4: number analyzed (Participants) | 15 | 15 | 17
  Adolescent - T4 | 11.80 (3.707) | 12.47 (2.722) | 9.41 (4.459)
  Adolescent - T5: number analyzed (Participants) | 12 | 14 | 15
  Adolescent - T5 | 11.92 (4.033) | 11.36 (2.590) | 11.80 (2.513)
Statistical Analysis 1: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares mothers in FBT to mothers in FBT+Parent-focused CRT; Test type: Superiority; p = .069, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 2: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares fathers in FBT to fathers in FBT+Parent-focused CRT; Test type: Superiority; p = .323, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 3: Comparison: Family Based Treatment (FBT) vs FBT w/Adolescent-focused Cognitive Remediation Therapy; This analysis compares adolescents in FBT to adolescents in FBT+Adolescent-focused CRT; Test type: Superiority; p = .225, generalized estimating equation

5. Primary Outcome: Change in Cognitive Flexibility - Verbal Fluency Switching of DKEFS
Description: The Delis Kaplan Executive Functioning System (D-KEFS) is a standardized assessment of executive functioning normed for ages 8-89 years of age. Raw scores are transformed to scaled scores: the mean is 10 with a standard deviation of 3. Higher scores indicate better performance on the test. Specific sub-tests were chosen to assess inhibitory control and cognitive flexibility. The hypothesis is that Cognitive Remediation Therapy (CRT) will increase flexibility in participants. The D-KEFS was administered at baseline (T1), after 4 weeks (T2), approximately 9 weeks (T3), approximately 17 weeks (T4), and end of treatment (T5). The D-KEFS Verbal Fluency assesses the ability to shift between concepts. Switching Accuracy assesses the number of times an accurate switch between categories occurs.
Time Frame: 6 months of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Number analyzed (Participants) | 63 | 57 | 57
score on a scale
  Mother - T1: number analyzed (Participants) | 20 | 19 | 19
  Mother - T1 | 11.90 (3.567) | 11.68 (3.637) | 11.95 (4.183)
  Mother - T3: number analyzed (Participants) | 19 | 16 | 17
  Mother - T3 | 11.63 (2.929) | 11.56 (1.590) | 11.24 (2.166)
  Mother - T4: number analyzed (Participants) | 16 | 16 | 17
  Mother - T4 | 14.06 (3.043) | 12.63 (3.284) | 13.65 (3.968)
  Mother - T5: number analyzed (Participants) | 12 | 15 | 15
  Mother - T5 | 11.58 (1.975) | 12.07 (1.335) | 12.13 (1.356)
  Father - T1: number analyzed (Participants) | 21 | 19 | 18
  Father - T1 | 11.81 (3.628) | 10.37 (3.890) | 11.50 (2.854)
  Father - T3: number analyzed (Participants) | 19 | 16 | 18
  Father - T3 | 11.68 (3.528) | 11.13 (2.705) | 11.56 (2.549)
  Father - T4: number analyzed (Participants) | 14 | 16 | 16
  Father - T4 | 12.71 (4.286) | 12.06 (3.958) | 12.00 (3.386)
  Father - T5: number analyzed (Participants) | 11 | 14 | 15
  Father - T5 | 12.45 (2.911) | 11.21 (2.155) | 11.53 (1.846)
  Adolescent - T1: number analyzed (Participants) | 20 | 19 | 18
  Adolescent - T1 | 11.45 (3.634) | 11.95 (2.549) | 11.28 (2.321)
  Adolescent - T3: number analyzed (Participants) | 18 | 16 | 17
  Adolescent - T3 | 11.56 (1.617) | 12.19 (1.559) | 10.88 (2.233)
  Adolescent - T4: number analyzed (Participants) | 15 | 15 | 17
  Adolescent - T4 | 12.20 (3.299) | 12.13 (2.90) | 10.18 (4.261)
  Adolescent - T5: number analyzed (Participants) | 12 | 14 | 15
  Adolescent - T5 | 12.00 (1.758) | 12.00 (1.414) | 11.93 (1.486)
Statistical Analysis 1: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares mothers in FBT to mothers in FBT+Parent-focused CRT; Test type: Superiority; p = .196, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 2: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares fathers in FBT to fathers in FBT+Parent-focused CRT; Test type: Superiority; p = .812, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 3: Comparison: Family Based Treatment (FBT) vs FBT w/Adolescent-focused Cognitive Remediation Therapy; This analysis compares adolescents in FBT to adolescents in FBT+Adolescent-focused CRT; Test type: Superiority; p = .499, generalized estimating equation — a priori threshold for statistical significance = .15

6. Primary Outcome: Change in Cognitive Flexibility - Sorting Test Description of DKEFS
Description: The Delis Kaplan Executive Functioning System (D-KEFS) is a standardized assessment of executive functioning normed for ages 8-89 years of age. Raw scores are transformed to scaled scores: the mean is 10 with a standard deviation of 3. Higher scores indicate better performance on the test. Specific sub-tests were chosen to assess inhibitory control and cognitive flexibility. The hypothesis is that Cognitive Remediation Therapy (CRT) will increase flexibility in participants. The D-KEFS was administered at baseline (T1), after 4 weeks (T2), approximately 9 weeks (T3), approximately 17 weeks (T4), and end of treatment (T5). The Sorting Test assesses flexibility in thinking and problem solving.
Time Frame: 6 months of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Number analyzed (Participants) | 63 | 57 | 57
score on a scale
  Mother - T1: number analyzed (Participants) | 18 | 17 | 17
  Mother - T1 | 11.94 (3.334) | 11.47 (1.972) | 12.47 (1.700)
  Mother - T3: number analyzed (Participants) | 14 | 13 | 12
  Mother - T3 | 12.21 (2.119) | 12.38 (1.446) | 13.50 (2.680)
  Mother - T4: number analyzed (Participants) | 10 | 10 | 11
  Mother - T4 | 12.80 (1.814) | 14.00 (2.449) | 14.00 (1,673)
  Mother - T5: number analyzed (Participants) | 7 | 9 | 4
  Mother - T5 | 13.86 (1.464) | 13.22 (1.787) | 16.25 (1.258)
  Father - T1: number analyzed (Participants) | 20 | 17 | 17
  Father - T1 | 11.80 (2.331) | 12.94 (2.358) | 12.35 (2.290)
  Father - T3: number analyzed (Participants) | 13 | 13 | 12
  Father - T3 | 12.15 (2.478) | 13.85 (2.478) | 12.92 (1.676)
  Father - T4: number analyzed (Participants) | 10 | 10 | 11
  Father - T4 | 12.50 (2.224) | 14.00 (2.404) | 12.82 (2.136)
  Father - T5: number analyzed (Participants) | 6 | 10 | 6
  Father - T5 | 14.00 (1.789) | 14.60 (2.366) | 15.00 (1.414)
  Adolescent - T1: number analyzed (Participants) | 19 | 17 | 17
  Adolescent - T1 | 11.37 (2.712) | 11.65 (1.693) | 10.35 (2.737)
  Adolescent - T3: number analyzed (Participants) | 12 | 13 | 11
  Adolescent - T3 | 11.33 (2.229) | 11.54 (1.808) | 11.00 (2.793)
  Adolescent - T4: number analyzed (Participants) | 9 | 10 | 11
  Adolescent - T4 | 13.22 (1.856) | 12.20 (2.044) | 11.27 (1.902)
  Adolescent - T5: number analyzed (Participants) | 7 | 10 | 6
  Adolescent - T5 | 12.171 (.488) | 12.00 (2.582) | 11.17 (2.483)
Statistical Analysis 1: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares mothers in FBT to mothers in FBT+Parent-focused CRT; Test type: Superiority; p = .446, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 2: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares fathers in FBT to fathers in FBT+Parent-focused CRT; Test type: Superiority; p = .647, generalized estimating equation
Statistical Analysis 3: Comparison: Family Based Treatment (FBT) vs FBT w/Adolescent-focused Cognitive Remediation Therapy; This analysis compares adolescents in FBT to adolescents in FBT+Adolescent-focused CRT; Test type: Superiority; p = .765, generalized estimating equation — a priori threshold for statistical significance = .15

7. Primary Outcome: Change in Self-Reported Shifting - BRIEF
Description: The Behavior Rating Inventory of Executive Functioning (BRIEF) is an ecologically valid clinical tool for measuring executive functioning across several domains in youth 5 to 18 years of age; the self-report version (BRIEF-2) was administered to adolescents. It has a comparable adult self-report version (BRIEF-A) normed for ages 18-90. Both versions of the BRIEF are normed by age and sex on a T-scale (mean = 50, SD = 10), and scores are considered clinically elevated if they are 65 or higher. Both have a number of clinical scales and indices. Lower scores indicate greater strengths in each area. The hypothesis is that Cognitive Remediation Therapy (CRT) will increase flexibility in participants, thus, we expect a reduction in scores for those in the CRT conditions. The BRIEF was administered at baseline (T1), after 4 weeks (T2), approximately 9 weeks (T3), approximately 17 weeks (T4), and end of treatment (T5). The BRIEF Shift assesses behavioral flexibility.
Time Frame: 6 months of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Number analyzed (Participants) | 63 | 57 | 57
score on a scale
  Mother - T1: number analyzed (Participants) | 21 | 19 | 19
  Mother - T1 | 58.38 (6.953) | 53.21 (7.843) | 51.79 (9.920)
  Mother - T3: number analyzed (Participants) | 19 | 16 | 18
  Mother - T3 | 56.47 (8.650) | 56.31 (11.001) | 54.28 (11.509)
  Mother - T4: number analyzed (Participants) | 15 | 16 | 17
  Mother - T4 | 56.07 (9.996) | 55.75 (12.557) | 52.94 (11.771)
  Mother - T5: number analyzed (Participants) | 12 | 15 | 15
  Mother - T5 | 55.92 (8.361) | 55.67 (12.210) | 53.27 (11.823)
  Father - T1: number analyzed (Participants) | 21 | 19 | 19
  Father - T1 | 50.67 (11.625) | 59.58 (9.924) | 53.43 (9.300)
  Father - T3: number analyzed (Participants) | 18 | 16 | 16
  Father - T3 | 52.17 (11.658) | 59.69 (8.592) | 46.63 (7.940)
  Father - T4: number analyzed (Participants) | 14 | 16 | 16
  Father - T4 | 50.71 (9.980) | 59.25 (8.993) | 47.25 (8.103)
  Father - T5: number analyzed (Participants) | 11 | 15 | 15
  Father - T5 | 47.55 (7.381) | 57.13 (10.453) | 48.07 (8.681)
  Adolescent - T1: number analyzed (Participants) | 21 | 19 | 19
  Adolescent - T1 | 60.86 (9.926) | 55.58 (12.389) | 58.16 (10.399)
  Adolescent - T3: number analyzed (Participants) | 17 | 15 | 17
  Adolescent - T3 | 58.71 (12.494) | 55.13 (11.618) | 55.59 (11.571)
  Adolescent - T4: number analyzed (Participants) | 14 | 16 | 17
  Adolescent - T4 | 60.36 (12.125) | 52.50 (11.770) | 54.82 (12.812)
  Adolescent - T5: number analyzed (Participants) | 11 | 13 | 15
  Adolescent - T5 | 58.18 (10.226) | 50.38 (9.726) | 54.87 (10.789)
Statistical Analysis 1: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares mothers in FBT to mothers in FBT+Parent-focused CRT; Test type: Superiority; p = .425, generalized estimating equation — a priori threshold for statistical significance = .15
Statistical Analysis 2: Comparison: Family Based Treatment (FBT) vs FBT w/ Parent-focused Cognitive Remediation Therapy; This analysis compares fathers in FBT to fathers in FBT+Parent-focused CRT; Test type: Superiority; p = .630, generalized estimating equation
Statistical Analysis 3: Comparison: Family Based Treatment (FBT) vs FBT w/Adolescent-focused Cognitive Remediation Therapy; This analysis compares adolescents in FBT to adolescents in FBT+Adolescent-focused CRT; Test type: Superiority; p = .854, generalized estimating equation — a priori threshold for statistical significance = .15

8. Primary Outcome: Dose of CRT
Description: Number of sessions necessary in order to change cognitive flexibility. This is the number of sessions needed for change to occur in cognitive flexibility. It is only calculated for the participants who received CRT and who had a significant change in flexibility above what was observed in FBT.
Time Frame: 6 months of treatment
Population: As parents did not hit a-priori milestones, we only calculated the number (count) of sessions needed for adolescents to have measurable improvement in cognitive flexibility.
Measure: Number; unit: Number of sessions
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
Number analyzed (Participants) | 21 | 0 | 19
Number of sessions | 0 |  | 8

ADVERSE EVENTS:
Time Frame: 6 months (from baseline intake to end of treatment)
Description: Definitions used for adverse events are the same as those used by clinicaltrials.gov.
Arm/Group | Family Based Treatment (FBT) | FBT w/ Parent-focused Cognitive Remediation Therapy | FBT w/Adolescent-focused Cognitive Remediation Therapy
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/63 | 1/57 | 0/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family Based Treatment (FBT) (N=63) | FBT w/ Parent-focused Cognitive Remediation Therapy (N=57) | FBT w/Adolescent-focused Cognitive Remediation Therapy (N=57)
Other (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — 1 adolescent presented to the hospital ED with chest pains originally thought not to be related to malnutrition that is a consequence of AN. Upon evaluation, the symptoms were determined to be due to malnutrition in the context of anorexia nervosa

LIMITATIONS AND CAVEATS:
The onset of the pandemic required that much data collection occur remotely, therefore, there is substantial missing data for Card Sort and Trail Making Test of the DKEFS. There were covid related delays in data scoring and analysis.

For each condition, we have a group of mothers, fathers, and youth. Each group is analyzed separately in each condition. We compared youth in FBT to youth in CRTA and parents in FBT to parents in CRTP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03928028/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03928028/ICF_000.pdf